CLINICAL TRIAL: NCT05432089
Title: The Effects of Oxytocin Administration to Patients and Therapists on Physiological Synchronization: a Randomized Controlled Pilot Study
Brief Title: The Effects of Oxytocin Administration to Patients and Therapists on Physiological Synchronization
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0002-22-SHA
Record Dates: First submitted 2022-06-16; First posted 2022-06-27 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Severe Mental Illness
Keywords: Oxytocin; Physiological Synchronization; Psychotherapy
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Drug: Intranasal Oxytocin
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Intranasal Oxytocin

INTERVENTIONS:
Drug: Intranasal Oxytocin — 24IU (12IU*2) of OT, Sorbitol, Benzyl, alcohol glycerol, distilled water.

SUMMARY:
Introduction: Oxytocin (OT) is a nine-amino acid neuropeptide, known to have a fundamental role in social communication. In a recent randomized, double-blind, placebo-controlled study carried out in Shalvata Mental Health Center, OT was administrated to patients suffering from severe mental health illness. The results indicated that OT has a clear beneficial effect on therapeutic outcomes. However, to our knowledge, the effect of OT administration to both patients and therapists on the therapeutic process was never tested. Substance administration to caregivers is therefore possible, and could, in some cases, provide further knowledge about the caregiving dynamics. Since we know the therapist's characteristics effect the therapeutic alliance and that OT is associated with the therapeutic alliance, patient-therapist bond, and therapy outcome, we are led to ask if OT administration to patients and therapists could allow for a deeper understanding of OT's effects on the therapeutic process.

Another variable found to be associated with the therapeutic process is Physiological Synchronization. Physiological Synchronization (PS) is a primarily interpersonal phenomenon which includes coordination of physiological signals between two or more interacting individuals. Despite the rising number of studies examining PS, its physiological and psychological mechanisms are yet to be fully understood. Based on literature indicating associations between OT and PS, and associations each of them has with the therapeutic process and its facilitators, in this study we wish to examine the influence of OT on PS through intranasal OT administration to patients alone and to patients and therapists together.

Research Hypotheses:

1. Patients receiving OT will demonstrate higher levels of PS during the measured session compared to patients receiving placebo.
2. Patients receiving OT will report higher levels of perceived therapist empathy as compared to patients receiving placebo.
3. These associations will be stronger when both patient and therapist receive OT in comparison to patient alone.
4. Changed in PS and empathy will be associated with OT even after controlling for patient rated alliance and session impact.
5. These findings will sustain after controlling for severity of symptoms and attachment patterns.

Method:

Participants. Sixty patients and their therapists will be recruited for the pilot study. Patients will be recruited from the inpatient adult psychiatric wards at Shalvata Mental Health Center. Therapists in this study will be comprised of psychologists, psychiatrists, and social workers, in different stages of seniority and training.

Instruments. Attachment patterns, symptom severity, side effects and therapeutic process measurements - working alliance, perceived empathy and session impact - will be assessed using self-report questionnaires. PS will be measured by recordings of the electrodermal activity (EDA) measured by skin conductance signals, using a galvanic skin response (GSR) device. Oxytocin Administration will be performed intranasally using a spray containing 24U.

Procedure. Sixty patients meeting inclusion criteria and their therapists will be recruited for the pilot study. Dyads will be randomized and double-blindly allocated to receive intra-nasal oxytocin or placebo. Dyads will be followed for two consecutive sessions, approximately at their fourth and fifth sessions. After signing informed consent forms, patients and therapists will complete therapeutic process measurements, and patients will be assessed for the severity of their symptoms and attachment patterns. Prior to the first session, patients will be administrated with either IN-OT or PLC and will wait for 30 minutes before the beginning of the session. Skin conductance synchrony will be measured during the session. At the end of the session, therapeutic process measurements will be assessed in both patients and therapists, and patients will complete a side-effect questionnaire. Prior to the second session, both patients and therapists will receive either IN-OT or PLC (each dyad will receive the same substance) and will wait for 30 minutes before the beginning of the session. Skin conductance synchrony will then be measured during the session. At the end of the session, therapeutic process measurements will be assessed in both patients and therapists alongside with a side-effect questionnaire.

The uniqueness of the proposed study is rooted in the view of the psychotherapy dyad as undetached, by focusing on the dyad and not on the patient alone. Focusing on patient-therapist synchronization lies on the understanding of the patient-therapist bond as co-dependent and co-affected. Such research could increase our understanding of PS between patient and therapist and its meaning in psychotherapy research and practice.

DETAILED DESCRIPTION:
Oxytocin (OT) is a nine-amino acid neuropeptide, known to have a fundamental role in social communication. Studies have shown that OT is involved in the attachment system in mammals and in mother-infant bond. Furthermore, studies demonstrate that OT enhances the ability to trust and improves the positive effects of social support during stress. In romantic relationships, OT was found to increase positive communication during conflictual discourse between partners, and was also found to be associated with different affiliative processes, such as empathy, emotional regulation, pro-social behavior, and sense of belonging.

In a recent randomized, double-blind, placebo-controlled study carried out in Shalvata Mental Health Center, OT was administrated to patients suffering from severe mental health illness. The results indicated that OT has a clear beneficial effect on therapeutic outcomes. However, to our knowledge, the effect of OT administration to both patients and therapists on the therapeutic process was never tested. Several studies have examined the influence of different types of substances on caretakers. For example, Modafinil administration was found to improved cognitive performance of emergency physicians following overnight shifts. Another study tested the influence of melatonin administration to emergency physicians working nightshifts and found a modest improvement in their day sleep and night alertness. Substance administration to caregivers is therefore possible, and could, in some cases, provide further knowledge about the caregiving dynamics. Since we know the therapist's characteristics effect the therapeutic alliance and that OT is associated with the therapeutic alliance, patient-therapist bond, and therapy outcome, we are led to ask if OT administration to patients and therapists could allow for a deeper understanding of OT's effects on the therapeutic process.

Another variable found to be associated with the therapeutic process is Physiological Synchronization. Physiological Synchronization (PS) is a primarily interpersonal phenomenon which includes coordination of physiological signals between two or more interacting individuals. In other words, PS involves two individuals or more who mutually impact one another to the point of synchronizing, without necessary physical or visual contact. It has been suggested that PS originates during intra-uterine life between mother and fetus and to maintain through the entire human lifespan. Despite the rising number of studies examining PS, its physiological and psychological mechanisms are yet to be fully understood. Recently, Feldman (2020) has offered a model linking synchronized behavior, affiliative processes, and OT, arguing that these three components function in the service of a superordinate meaning system responsible for Human Resilience. However, to the best of our knowledge, the hypothesis of OT as the mediating neuro-hormone of PS is yet to be tested.

Based on literature indicating associations between OT and PS, and associations each of them has with the therapeutic process and its facilitators, in this study we wish to examine the influence of OT on PS through intranasal OT administration to patients alone and to patients and therapists together.

Research Hypotheses

1. Patients receiving OT will demonstrate higher levels of PS during the measured session compared to patients receiving placebo.
2. Patients receiving OT will report higher levels of perceived therapist empathy as compared to patients receiving placebo.
3. These associations will be stronger when both patient and therapist receive OT in comparison to patient alone.
4. Changed in PS and empathy will be associated with OT even after controlling for patient rated alliance and session impact.
5. These findings will sustain after controlling for severity of symptoms and attachment patterns.

Importance of the study The uniqueness of the proposed study is rooted in the view of the psychotherapy dyad as undetached, by focusing on the dyad and not on the patient alone. Focusing on patient-therapist synchronization lies on the understanding of the patient-therapist bond as co-dependent and co-affected. Such research could increase our understanding of PS between patient and therapist and its meaning in psychotherapy research and practice. Furthermore, the implications of such study could facilitate the understanding of the mechanisms of change in psychotherapy in a way that could be manipulated in the future.

Method Participants Sixty patients and their therapists will be recruited for the pilot study. Patients will be recruited from the inpatient adult psychiatric wards at Shalvata Mental Health Center. Inclusion criteria is: (a) age above 18. (b) any type of psychiatric illness. (c) hospitalization in one of the inpatients wards. Patients will be excluded from the research if they (a) are going through a severe psychotic episode, or (b) if pregnant according to self-report. Therapists in this study will be comprised of psychologists, psychiatrists, and social workers, in different stages of seniority and training. Therapists will be excluded from the study if pregnant according to self-report.

Instruments Attachment and outcome measurements are assessed for statistical control, and the therapeutic process measurements - therapeutic alliance, perceived empathy and session impact - are the dependent variables.

The Hopkins Symptom Checklist. A self-report questionnaire measuring symptoms of depression and anxiety. The HSCL-11 is a brief version of the SCL-90-R and it includes 11 items assessing symptomatic distress. The HSCL-11 is highly correlated with the Global Severity Index (r = .91) and has high internal consistency. The measure will be utilized at baseline to assess baseline levels of distress.

The Experience in Close Relationship Scale (ECR). A self-report questionnaire evaluating anxious and avoidant attachment in adults. It consists of 36 items divided to two dimensions: 18 items reflecting anxious attachment, while the other 18 items reflecting avoidant attachment. Participants indicate the extent to which they agree/disagree with each item in terms their general experience of close relationships on a 7-point scale ranging from not at all (1) to very much (7). Reliability and validity of the ECR have been repeatedly demonstrated. The measure will be utilized at baseline to assess attachment patterns.

The Working Alliance Inventory - Short Revised (WAI - SR). A self-report questionnaire that aims to evaluate patient-therapist working alliance through three aspects: agreement on therapy goals, agreement on therapeutic tasks and patient-therapist positive emotional bond. The WAI-SR is a brief version of the original 36-item WAI, and an extended version of the 6-item Working Alliance Inventory (WAI-6). The WAI-SR consists of 12 items rated on a 6-point scale ranging from not at all (1) to very much (6). The questionnaire has two versions: one assessing the alliance from the patient's point of view and the other assessing it from the therapist's point of view. This measurement was translated to hebrew and has demonstrated excellent reliability, convergent validity, and predictive validity.

The Barrett-Lennard Relationship Inventory - Empathy Scale (BLRI). A self-report questionnaire that relies on Rogers' (1957) four essential components for the achievement of positive therapeutic change: empathic understanding, level of regard, unconditionality of regard and congruence. Together, these components form four sub-scales, each consists of 16 items, 64 items in total. For the porpuses of the current study, the empathy sub-scale will be utilized. The sub-scale consists of 16 items and is rated in a 6-point scale. The questionnaire has two versions: one measuring the perceived empathy of others towards me, which will be filled by the patient, and another measuring "my perceived empathy for others", which will be filled by the therapist. The measure was found highly reliable, with internal consistency of 0.91 for the entire questionnaire, and 0.83 for the empathy sub-scale.

Session Evaluation Questionnaire (SEQ). A self-report questionnaire assessing the effects of a psychotherapy session through different aspects of the patient's views and feelings regarding the session. It consists of a 7-point scale of 20 bipolar adjectives (for example - 1-"sad" ranging to 7-"happy"). The adjectives refer to two dimensions: session (for example - "the current session was…") and post-session (for example - "now I'm feeling…"). The SEQ is divided to four sub-scales of session and post-session: depth, flow, awareness and positivity. The depth sub-scale measures perceived efficacy and value of the session; the flow sub-scale measures perception of comfortability, calmness and peacefulness of the session; the awareness sub-scale measures the extent of energetic feeling post-session; the positiveness sub-scale measures the extent of positive feeling post-session. The SEQ demonstrated high internal consistency (α = .90) alongside high validity.

Side-effects questionnaire. A self-report scale aimed to assess potential side effects of IN-OT based on reports from past studies. It consists of 18 usual and unusual possible treatment side-effects. The questionnaire was constructed in order to provide indications of side-effects which might warrant additional safety considerations.

Electrodermal Activity (EDA). PS will be measured by the recordings of the electrodermal activity (EDA) signals using a galvanic skin response (GSR) device. The GSR device requires the attachment of two wireless electrodes to the subject's fingers. EDA was chosen due to recent developed analytic approaches for computing and interpretating PS processes based on EDA data. The AMIco algorithm identifies the picks and valleys in the EDA curves of the patient and therapist and tests their compatibility. The algorithm maximizes the probability of EDA correlation identification.

Oxytocin Administration. Intra-nasal OT (IN-OT) will be performed using a spray containing 24IU (12IU administered to each nostril), sorbitol, benzyl, alcohol glycerol, distilled water. Control group (PLC) will be administered using the same spray, containing the same components but the OT. Dosage and administration method was determined by standard OT studies guidelines. The two substances will be prepared immediately after randomization by an external trained nurse who has no relations to the study. The nursing staff will administer the substance after proper training by the chief hospital pharmacist and principal investigator.

Procedure Sixty patients meeting inclusion criteria and their therapists will be recruited for the pilot study. Dyads will be randomized and double-blindly allocated to receive intra-nasal oxytocin or placebo. Dyads will be followed for two consecutive sessions, approximately at their fourth and fifth sessions. After signing informed consent forms, patients and therapists will complete therapeutic process measurements, and patients will be assessed for the severity of their symptoms and attachment patterns. Prior to the first session, patients will be administrated with either IN-OT or PLC and will wait for 30 minutes before the beginning of the session. Skin conductance synchrony will be measured during the session. At the end of the session, therapeutic process measurements will be assessed in both patients and therapists, and patients will complete a side-effect questionnaire. Prior to the second session, both patients and therapists will receive either IN-OT or PLC (each dyad will receive the same substance) and will wait for 30 minutes before the beginning of the session. Skin conductance synchrony will then be measured during the session. At the end of the session, therapeutic process measurements will be assessed in both patients and therapists alongside with a side-effect questionnaire.

Patient safety and study ethics Studies have shown that OT administration has very low potential side-effects. 5-6% of the subjects reported an increase in calmness and euphoria sensations, lightheadedness and a headache, while 3% of the subjects reported stimulated nostrils resulting from the spray administration and dry mouth. Importantly, previous studies gave evidence that OT does not harm the effectiveness of standard antidepressant medication. To ensure optimal safety, the side effects profile will be evaluated throughout the intervention period by the treating psychiatrist, and participation will be ceased if needed.

Ethically, participants will be well informed of the possibility to drop out from the study at any time. Additionally, patients will be informed that dropping out will not affect the treatment they are receiving, and that the information gathered from them will not be accessible to their therapists.

Statistical Strategy To provide initial assessment of IN-OT's effectivity compared to PLC, we will perform a comparison between the clinical courses of each dyad, using Jacobson and Truax (1991) approach for Reliable Clinical Change (index). Cohen's d will be used for effects sizes. Differences in effectivity will be demonstrated in Cramer's V, as indicators for effects sizes. Physiological Synchronization will be assessed using Truth and Bias models. All statistical analysis will be performed using SPSS software and R software.

ELIGIBILITY:
Patients Inclusion Criteria:

* age above 18.
* any type of psychiatric illness.
* hospitalization in one of the inpatients wards.

Patients Exclusion Criteria:

* current severe psychotic episode
* pregnancy according to self-report.

Therapist Inclusion Criteria:

* psychologists, psychiatrists, and social workers, in different stages of seniority and training.

Therapist Exclusion Criteria:

* pregnancy according to self-report.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
skin conductance synchrony | 1-2 weeks including 2 consecutive psychotherapy sessions
  as measured by GSR devices during sessions

SECONDARY OUTCOMES:
working alliance | 1-2 weeks including 3 measurements: baseline, post-session 1 and post-session 2.
  as measured by The Working Alliance Inventory - Short Revised (WAI - SR; Hatcher & Gillapsy, 2006).
perceived empathic understanding | 1-2 weeks including 3 measurements: baseline, post-session 1 and post-session 2.
  as measured by The Barrett-Lennard Relationship Inventory - Empathy Scale (BLRI; Barrett-Lennard, 1962).
session impact | 1-2 weeks including 2 measurements: post-session 1 and post-session 2.
  as measured by the Session Evaluation Questionnaire (SEQ; Stiles & Snow, 1984).

CONTACTS AND LOCATIONS:
Locations (1):
- Shalvata Mental health Center, Hod HaSharon, Israel